CLINICAL TRIAL: NCT01879657
Title: An Open-label, Single-dose, Clinical Trial of 68Ga-DOTATATE (GalioMedix™) PET-CT Scan for Diagnosis of Primary and Metastatic Somatostatin Receptor-positive Neuroendocrine Tumors (NETs)
Brief Title: 68Ga-DOTATATE PET-CT for Diagnosis of Neuroendocrine Tumors (NETs)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radio Isotope Therapy of America (Other)
Collaborators: Radiomedix, Inc. (Industry); Excel Diagnostics and Nuclear Oncology Center (Other)
Responsible Party: Principal Investigator, Ebrahim Delpassand, President, Radio Isotope Therapy of America
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 117289
Record Dates: First submitted 2013-04-11; First posted 2013-06-18 (Estimated); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Neuroendocrine Carcinoma
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — gallium Ga 68 dotatate; Positron Emission Tomography Computed Tomography; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 68Ga-DOTATATE (Experimental): All participants will be injected with 68Ga-DOTATATE approximately 60 minutes before PET/CT scan.
  Interventions: Drug: 68Ga-DOTATATE; Diagnostic Test: PET/CT; Diagnostic Test: 111In-pentetreotide OctreoScan; Diagnostic Test: MRI

INTERVENTIONS:
Drug: 68Ga-DOTATATE — 68Ga-DOTATATE (3-5 mCi ±25%; 111-185 MBq) is administered as a single intravenous bolus injection in each participant. These injections were performed within 28 days after the Octreoscan.
  Other Names: Gallium-68 DOTATATE; [⁶⁸Ga]-DOTA-Tyr3-Octreotate; 68Ga DOTA-TATE
Diagnostic Test: PET/CT — 68Ga-DOTATATE PET images will be acquired 60 ±30 minutes after injection of 68Ga-DOTATATE. 68Ga-DOTATATE PET images were performed within 28 days after the Octreoscan.
  Other Names: PET-CT Scan
Diagnostic Test: 111In-pentetreotide OctreoScan — OctreoScan™ was performed after intravenous injection of 111In-pentetreotide, a radiopharmaceutical that binds to somatostatin receptors, if the patient had not undergone such imaging as a standard of care. Subsequent planar and/or SPECT imaging was used to detect somatostatin receptor-positive lesions.
Diagnostic Test: MRI — MRI (Standard of Care)
  Other Names: Magnetic Resonance Imaging (MRI)

SUMMARY:
To evaluate the concordance and discordance between results of 68Ga-DOTATATE PET-CT scan and OctreoScan ® which is considered standard of care diagnostic test for neuroendocrine cancers and other imaging modalities like CT scan/MRI as gold standard.

DETAILED DESCRIPTION:
The number of lesions that could be identified clearly as single foci will be determined for each patient. The same anatomic areas will be imaged with 68Ga-DOTATATE PET and 111In-penteoctreotide Scintigraphy to ensure relevant comparison of lesion detection. Because of confluence and inability to clearly delineate single liver lesions in some cases, liver metastases will be classified as 1 organ metastasis, independent of the number of liver metastases present. Lymph nodes smaller than 1 cm on CT or MRI and showing marked avidity for 68Ga- DOTATATE and 111In-penteoctreotide will be labeled as positive for disease. The presence of lesions will be confirmed by cross-sectional imaging of all patients with CT or MRI.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Subjects of either sex, aged ≥18 years
* Histologically and/or clinically confirmed and/or suspected NET and/or A diagnostic imaging study including but not limited to CT or MRI or FDG PET/CT, NaF PET/CT, bone scan, ultrasound, etc. of the tumor region or suspected area within the 4 weeks of dosing day
* Recent Blood test results (within 2-4 weeks predose) as WBC: ≥2 x 109/L, Haemoglobin: ≥8.0 g/dL, Platelets: ≥50 x 109/L, ALT, AST, AP:≤ 5 times ULN [ ULN for ALT, AST and AP is 70, 20 and 20 Units/I respectively], Bilirubin: ≤3 times ULN [ULN for total bilirubin is 1.3mg/dL]
* Serum creatinine: Serum creatinine: <170 μmol/L
* egative pregnancy test in women capable of child-bearing

Exclusion Criteria:

* Known hypersensitivity to DOTA, to 68Gallium, to Octreotate or to any of the excipients of 68Ga-DOTATATE
* Therapeutic use of any somatostatin analogue, including Sandostatin® LAR (within 28 days) and Sandostatin® (within 2 days) prior to study imaging. If a patient is on Sandostatin® LAR a wash-out phase of 28 days is required before the injection of the study drug
* Pregnant or breast-feeding women
* Current somatic or psychiatric disease/condition that may interfere with the objectives and assessments of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2017-12-05 (Actual)

PRIMARY OUTCOMES:
Number of lesions detected by 68GA-DOTATATE compared to conventional imaging technique | SOT within 28 days before 68Ga-DOTATATE PET/CT scan
  We want to determine if the 68Ga-DOTATATE PET/CT scan changes care plans compared to conventional imaging/diagnostic techniques (Octreoscan, MRI).

SECONDARY OUTCOMES:
Frequency and severity of Adverse Events | 4 days
  Adverse events will be collected from the time of 68Ga-DOTATATE injection until 48 hours post-injection visit. Adverse events will be classified using criteria for adverse events (CTCAE) Version 4.

CONTACTS AND LOCATIONS:
Overall Officials: Ebrahim Delpassand, MD, Principal Investigator — Radiomedix, Inc.
Locations (1):
- Radio- Isotope Therapy of America, Houston, Texas, United States